CLINICAL TRIAL: NCT02211820
Title: PET Imaging in Chronic Traumatic Encephalopathy
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140164; 14-M-0164
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-10-12

CONDITIONS: Brain Disease; Brain Mapping
Keywords: Encephalopathy; Imaging Studies; Dementia; Cerebellar Cortical Atrophy
MeSH Terms: conditions — Brain Diseases; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Chronic traumatic encephalopathy (CTE) is a brain disease caused in part by head injury. The brain changes from CTE can only be seen at autopsy. Researchers want to test a new brain scan to help diagnose CTE in living patients.

Objective:

- To determine if a new type of brain scan can detect changes that occur in chronic traumatic encephalopathy.

Eligibility:

- Adults age 18 60 with previous head injury or participation in certain sports.

Design:

* Participants will be screened with:
* Physical exam
* Blood and urine tests
* Tests of thinking, mood, and memory
* 30-minute magnetic resonance imaging (MRI) brain scan. A magnetic field and radio waves take pictures of the brain. Participants will lie on a table that slides into a metal cylinder. They will get earplugs for the loud knocking sounds.
* Visit 1: Participants will have a 70-minute PET scan of the brain with a small amount of a radioactive chemical. That will be injected through an intravenous tube (catheter) in each arm. A catheter will also be put into an artery at the wrist or elbow.
* Participants will lie on a bed that slides in and out of a donut-shaped scanner. A plastic mask may be molded to their face and head. Vital signs and heart activity will be checked before and during the scan.
* Blood and urine will be taken before and after the scan.
* Participants will be checked on by phone the next day.
* Visit 2: Participants will repeat Visit 1 with a different chemical and no artery catheter.
* Visit 3: Participants may have a spinal tap. Some fluid will be removed by needle between the bones in the back.

DETAILED DESCRIPTION:
Objective: To determine if the PET radioligand [11C]PBB3 can detect aggregates of tau protein in the brains of patients with history of traumatic brain injury (TBI) and suspected chronic traumatic encephalopathy (CTE).

Study population: The proposed study will include 40 subjects. Twenty will be patients with history of TBI and suspected CTE and 20 will be healthy cognitively normal volunteers without history of TBI.

Design: Subjects will undergo medical screening and have brain MRI and neuropsychological testing performed. Subjects will undergo one brain PET scan with [11C]PBB3 to detect aggregates of tau protein. Subjects will also have one brain PET scan with [11C]Pittsburgh compound B (PIB) to detect amyloid plaques. Subjects will be asked to have a lumbar puncture to measure CSF tau concentrations.

Outcome measures: The primary outcome measure will be the amount of [11C]PBB3 binding in the brain. We will quantify the radioligand s brain uptake, washout, plasma clearance, and distribution volume using compartmental modeling. Distribution volume of [11C]PBB3 is proportional to the density of insoluble paired helical filaments of tau and is equal to the ratio at equilibrium of uptake in brain to the concentration of parent radiotracer in plasma. As an exploratory measure, we will determine if there is a relationship between [11C]PBB3 binding in brain and gray matter loss on MRI. We will also measure the amount of [11C]PIB binding in the brain using the Logan reference tissue method with cerebellum as reference.

ELIGIBILITY:
* INCLUSION CRITERIA:<TAB>

<TAB>

* For patients:

  * History of head injury resulting from past or current participation in one or more contact sports (hockey, football, or boxing). Patients may have history of structural brain injury (i.e., injury accompanying abnormality on MRI or CT scan), concussion without structural injury (mild TBI), or repetitive sub-concussive injury.
  * Meets DMS-V criteria for Major Neurocognitive Disorder or Mild Neurocognitive Disorder
  * Age 18 to 60 years.
  * Ambulatory.
  * Patients unable to provide informed consent must have a surrogate decision maker.
* For healthy controls:

  * Healthy without past or present history of brain disease.
  * Age 18 to 60 years.
  * Able to provide informed consent.

EXCLUSION CRITERIA:

* Past or present history of a brain disorder other than TBI.
* For patients: Subjects with abnormal brain imaging findings that suggest a diagnosis other than TBI or a second lesion such as brain tumor in addition to the changes consistent with TBI.
* For controls: past or present history of either a single concussion or more severe TBI, or of repetitive sub-concussive injury due to contact sport participation.
* Serious medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries. The Principal Investigator of this protocol will determine whether the subject needs to be excluded.
* The DSM-V criteria for Major Neurocognitive Disorder are as follows:

  --Evidence of significant cognitive decline from a previous level of performance in one or more cognitive domains (complex attention, executive function, learning and memory, perceptual-motor, or social cognition) based on:
  * Concern of the individual, a knowledgeable informant, of the clinician that there has been a significant decline in cognitive function.
  * A substantial impairment in cognitive performance, preferably documented by standardized neuropsychological testing, or, in its absence, another qualified clinical assessment.
* The cognitive deficits interfere with independence in everyday activities (i.e. at a minimum, requiring assistance with complex instrumental activities of daily living such as paying bills or managing medications)
* The cognitive deficits do not occur exclusively in the context of delirium.
* The cognitive disorder is not better explained by another mental disorder (e.g. major depressive disorder, schizophrenia).
* Criteria for Mild Neurocognitive Disorder are as follows:

  * There is evidence of modest cognitive decline from a previous level of performance in one or more of the domains outlined above based on:

    * Concern of the individual, a knowledgeable informant, or the clinician.
    * Decline in neurocognitive performance, preferably documented by standardized neuropsychological testing, or, in its absence, another qualified clinical assessment.
  * The cognitive deficits are insufficient to interfere with independence (eg, instrumental activities of daily living, like more complex tasks such as paying bills or managing medications,

are preserved), but greater effort, compensatory strategies, or accommodation may be required to maintain independence.

* The cognitive deficits do not occur exclusively in the context of a delirium.
* The cognitive deficits are not primarily attributable to another mental disorder (eg, major depressive disorder, schizophrenia).

There are no restrictions on medications. Since disease modifying therapy for tauopathies (including CTE and Alzheimer s disease) do not currently exist, no currently available medications, either prescribed or over-the-counter, are expected to confound the results of this study. Anti-inflammatory medications, including NSAIDs, are not expected to significantly reduce tau aggregation in CTE patients, based on the failure of these medications to prevent disease progression in Alzheimer s disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-08-01; Primary Completion 2016-06-20 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Amount of 11C-PBB3 binding in brain as measured with PET | 1 year

SECONDARY OUTCOMES:
Amount of brain atrophy as measured with MRI.Amount of 11C-PIB binding in brain as measured with PET | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baugh CM, Stamm JM, Riley DO, Gavett BE, Shenton ME, Lin A, Nowinski CJ, Cantu RC, McKee AC, Stern RA. Chronic traumatic encephalopathy: neurodegeneration following repetitive concussive and subconcussive brain trauma. Brain Imaging Behav. 2012 Jun;6(2):244-54. doi: 10.1007/s11682-012-9164-5. PMID 22552850
- [Background] Braskie MN, Klunder AD, Hayashi KM, Protas H, Kepe V, Miller KJ, Huang SC, Barrio JR, Ercoli LM, Siddarth P, Satyamurthy N, Liu J, Toga AW, Bookheimer SY, Small GW, Thompson PM. Plaque and tangle imaging and cognition in normal aging and Alzheimer's disease. Neurobiol Aging. 2010 Oct;31(10):1669-78. doi: 10.1016/j.neurobiolaging.2008.09.012. Epub 2008 Nov 11. PMID 19004525
- [Background] Chien DT, Bahri S, Szardenings AK, Walsh JC, Mu F, Su MY, Shankle WR, Elizarov A, Kolb HC. Early clinical PET imaging results with the novel PHF-tau radioligand [F-18]-T807. J Alzheimers Dis. 2013;34(2):457-68. doi: 10.3233/JAD-122059. PMID 23234879